CLINICAL TRIAL: NCT03904264
Title: Feasibility and Acceptability of Using Low-Gain Hearing Aids for Bothersome Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C3196-P
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Tinnitus; Hearing Aids; Normal Hearing
Keywords: tinnitus; hearing aids; normal hearing
MeSH Terms: conditions — Tinnitus | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: For this pilot study 20 eligible adults with bothersome tinnitus and normal hearing thresholds from audiometric frequencies .25 kHz through 4 kHz will be provided with hearing aids. Eligible adults with tinnitus and normal hearing are the only participants for whom an intervention will be provided as part of the study. Fifteen VA clinical audiologists will be interviewed to document opinions, procedures, and rationale used clinically to make decisions regarding fitting mild amplification for tinnitus on Veterans with bothersome tinnitus and normal hearing thresholds. No intervention will be provided to the participating audiologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hearing Aid Study (Experimental): Measure the reduction in tinnitus handicap when mild amplification through receiver-in-the-canal hearing aids is provided to adults with bothersome tinnitus and normal hearing thresholds.
  Interventions: Device: Receiver in the canal (RIC) hearing aids
- VA Clinician Interviews (No Intervention): Document the opinions, procedures, and rationale used clinically to make decisions regarding fitting mild amplification for tinnitus on Veterans with bothersome tinnitus and normal hearing thresholds. The data for this arm of the study will be collected via telephone interview.

INTERVENTIONS:
Device: Receiver in the canal (RIC) hearing aids — The RIC hearing aids fitted to subjects in arm 1 of the study will be manufactured by Widex.
  Arms: Hearing Aid Study

SUMMARY:
Tinnitus - defined as ringing, humming, or other sounds in the ears or head - is a very common problem for Veterans. Hearing aids that deliver low-level amplification are being used by audiologists to help people with tinnitus who also have normal hearing. However, there is a lack of research evidence showing that this practice is effective. Despite this fact, the practice clearly is spreading. Reports from audiologists in the field as well as research presentations refer to hearing aids being used in this way. Use of hearing aids has been shown to reduce distress from tinnitus for people with hearing loss. Additionally, the use of external sound to help reduce the impact of tinnitus has been shown to be effective. There is clearly a gap in the research regarding the use of hearing aids as a therapeutic method to manage tinnitus when hearing is considered normal. This study will obtain pilot data evaluating people with normal hearing and bothersome tinnitus to find out whether low-level amplification through hearing aids may provide benefit.

DETAILED DESCRIPTION:
Tinnitus - defined as ringing, humming, or other sounds in the ears or head - is the most prevalent service-connected disability among Veterans. Tinnitus affects 10-15% of the adult population. For about 20% of these, tinnitus impacts their lives with respect to sleep disturbance, impaired concentration, and/or emotional reactions. These 20% are the most in need of clinical services. It has been shown that providing amplification via hearing aids for people with hearing loss can also be beneficial in reducing functional effects of tinnitus, presumably because amplifying environmental sounds reduces the contrast between the tinnitus and background sound, allowing the tinnitus to be more easily ignored. There have been increasing reports from the field of audiologists providing hearing aids set to deliver low-gain amplification on patients with bothersome tinnitus who are not otherwise hearing aid candidates, with beneficial outcomes. However, this nontraditional fitting practice has not been formally evaluated, so there is no research evidence to support the practice. It is essential for VA to show evidence supporting such practices to justify the use (and expense) of these devices with patients who otherwise do not qualify to receive hearing aids.

The proposed project is a pilot study that would lay the groundwork for a future full randomized controlled trial (RCT) evaluating the use of low-gain amplification for bothersome tinnitus in patients with normal hearing. A pilot sample of 20 Veterans with normal hearing thresholds and bothersome tinnitus will be fit with mild amplification through receiver-in-the-canal hearing aids. Hearing aids will be programmed to provide a low-level of amplification, using NAL-NL2 guidelines for target gain. Outcome measures will be evaluated pre-fit and post-fit at two follow-up time points (2 weeks and 3 months post-fit). Outcomes will include the Tinnitus Functional Index (TFI), Hearing Handicap Inventory for Adults (HHIA) and the Quick Speech in Noise (QuickSIN) test. Outcomes pre and post hearing aid fit will be compared to evaluate whether the hearing aids provided benefit to participants in terms of their tinnitus and hearing outcomes. Additionally, participants will be interviewed at their last visit to find out their self-reported benefit from the hearing aids, as well as any barriers they encountered to wearing the hearing aids.

Additionally, a group of VA clinical audiologists will be interviewed by telephone. These clinicians will be identified via an email survey sent to the VA audiologist email group, asking whether they are providing low-gain amplification for bothersome tinnitus to patients with normal hearing. The survey will also ask audiologists to volunteer if they are willing to participate in a brief telephone interview. The aim will be to identify at least ten audiologists who are fitting hearing aids in this way, and up to five who are not. These audiologists will be interviewed over the telephone to find out why they have incorporated this into their clinical practice (or why they have not), and inquire about specific fitting procedures and criteria for identifying candidates that they have used. These responses will inform the protocol of the future RCT.

At the conclusion of this project, enough information will be collected to propose a controlled study of low-gain amplification for bothersome tinnitus in people with normal hearing. The protocol for that project will be informed by both the successful aspects of the pilot protocol as well as the input from VA clinicians who are doing this in the field. A preliminary evaluation of benefit provided by these hearing aids will provide justification for a large controlled study. Finally, the pilot data will provide the basis for a power calculation to determine sample size, as well as an estimate of drop-out rate to sufficiently adjust for attrition. A full RCT demonstrating efficacy of low-gain amplification for bothersome tinnitus in people with normal hearing would provide needed evidence supporting a clinical practice that has already gained some traction both within and outside VA. Robust research evidence is needed to support the continuation and future expansion of this practice.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the Hearing Aid study include:

* a score of 5 or greater on section A the Tinnitus and Hearing Survey during the telephone screening; and
* air conduction hearing thresholds of 25 dB HL or better from .25 kHz through 4 kHz bilaterally as measured at the first study visit;
* must not be a current hearing aid user; and
* capable of consenting and participating (including ability to communicate in English).

Inclusion criteria for the VA Clinician Interviews:

-simply VA audiologists willing to participate.

Exclusion Criteria:

Exclusion criteria for the Hearing Aid study include:

* an air conduction hearing threshold greater than 25 dB HL from .25 kHz through 4 kHz;
* significant conductive hearing loss-defined as an air-bone gap of 15 dB at more than two frequencies in one ear, or an air-bone gap greater than 20 dB at any one frequency;
* suspicion of secondary (somatic) tinnitus, or Meniere's disease (either of which can be ruled out with an examination by an appropriate physician);
* currently a hearing aid user; or
* any mental, emotional, or health conditions that would preclude full study participation.

Exclusion criteria for the VA Clinician Interviews are:

* not an audiologist
* not a VA employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Zaugg, AuD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hearing Aid Study | VA Clinician Interviews
Started | 11 | 54
Completed | 3 | 17
Not Completed | 8 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hearing Aid Study | VA Clinician Interviews | Total
Number analyzed (Participants) | 11 | 54 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data was not collected for the interviews
  Years
    number analyzed (Participants) | 11 | 0 | 11
    (all) | 41.45 (8.69) |  | 41.45 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was not collected for interviews
  Participants
    number analyzed (Participants) | 11 | 0 | 11
    Female | 2 | 0 | 2
    Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data was not collected for interviews
  Participants
    number analyzed (Participants) | 11 | 0 | 11
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 11 | 0 | 11
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data was not collected for interviews
  Participants
    number analyzed (Participants) | 11 | 0 | 11
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 9 | 0 | 9
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 54 | 65

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index Change
Description: The Tinnitus Functional Index (TFI) is a statistically validated measure of the functional impact of tinnitus. The TFI was developed to be sensitive to changes in function as a result of intervention for tinnitus. Range is 0 - 100, higher numbers indicates greater level of distress and functional impact.
Time Frame: The Tinnitus Functional index will be administered at baseline, 2-3 weeks after baseline, and 3 months after baseline
Population: TFI was not administered for VA Clinician Interviews
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hearing Aid Study
Number analyzed (Participants) | 11
units on a scale
  Baseline | 53.31 (22.68)
  2-3 weeks: number analyzed (Participants) | 8
  2-3 weeks | 44.10 (23.02)
  3 months: number analyzed (Participants) | 3
  3 months | 64.93 (25.25)

ADVERSE EVENTS:
Description: Adverse Events were not monitored for this study
Arm/Group | Hearing Aid Study | VA Clinician Interviews
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03904264/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT03904264/ICF_000.pdf